CLINICAL TRIAL: NCT04671654
Title: Systematic Evaluation of Human Explant Model Systems Engineering
Acronym: SEEDLING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Niels Halama, Head of Department Translational Immunotherapy DKFZ, University Hospital Heidelberg
Other Study IDs: U1111-1254-2831-S-507/2019; U1111-1254-2831 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-11-11; First posted 2020-12-17 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor, Adult
Keywords: cancer; metastases; immunotherapy; radiation; chemotherapy; targeted therapy
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Explant Models
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All current forms of therapy for tumor patients are essentially based on clinical, genomic or histopathological criteria for the choice of therapy. However, the change in the tissue during therapy is of particular importance for patients, both with regard to the development of resistance and the side effect profile. This applies in particular to immunotherapies and their use in advanced tumor diseases. Preliminary work on the fully human tumor explant model has shown that the use of human donor tissue in the context of a special bioreactor makes it possible to improve the possibilities of predicting and better understanding the mechanism of action of a therapeutic agent. Since there is a considerable need for personalized and thus improved therapy management in the field of oncology, the aim of this study is on the one hand to improve the decisive tissue parameters for the cultivation of human donated material and on the other hand to understand the basic reaction patterns of the tissue to therapies.

DETAILED DESCRIPTION:
Personalized therapy is still one of the great goals of oncology. In view of the success of checkpoint inhibitor therapies in selected solid tumors, the question remains why other tumor diseases do not respond in the same way to the therapy. However, this is not only limited to immunotherapies. In principle, the understanding of the dynamic changes in a patient's tissue has so far been very limited, both for predicting a therapy success and with regard to the mechanistic understanding of how a therapy works. Model systems for diseases are often animal models that reproduce the complexity of a multi-organ system, but show significant differences to humans at the tissue level and therefore have only little informative value. Cell culture experiments, on the other hand, have only little informative value with regard to the overall behavior of a tissue or even an organ or the disease situation. "Naturalistic" co-culture in the Petri dish (such as with organoid systems) does not allow any sensible transferable insights, even if complex cell compositions of fibroblasts, endothelium or immune cells are used. In contrast, there is another problem for in vivo tumor models: either there is a lack of flexibility with regard to the structural context or the species-specific system properties do not allow any conclusions to be drawn about the situation in humans. This is a massive limitation, especially for translational studies. The Tumor Explant Model System developed by us allows the structural integrity of the tissue context to be maintained in the context of obtaining a biopsy or removing a resection. The tissue sample obtained in this way is kept in equilibrium via a bioreactor and can thus be used for tests or is preserved in its context of the tissue. It is also possible in the sense of a personalized diagnosis and therapy to take into account the individual bandwidth of the composition of the tumor microenvironment. This approach has already been validated in a prospective study and the transferability of the results from the explant models to humans has been proven. In this situation, the systematic construction of explant models for other tumor entities and the use of these models for therapy development and for better understanding of pathoregulation in tissues. In addition to the tissue samples donated by the study participants, blood cells can also be used for testing the tissue.hand to understand the basic reaction patterns of the tissue to therapies.

ELIGIBILITY:
Inclusion Criteria:

* Tissue material for Explant Model generation available or accessible

Exclusion Criteria:

* curatively resected/treated tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with solid tumor diseases in a non-curative setting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Tissue Biopsy Specimen vs Tumor Explant Model Prediction | up to 24 weeks
  Comparison of serial biopsy measurements to Explant Model measurements in the context of individual Patient variability, Serial biopsy timepoints can vary between 1 day up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Jaeger, Prof. Dr. med., Study Chair — University Hospital Heidelberg
Locations (1):
- University of Heidelberg / NCT, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Halama N, Zoernig I, Berthel A, Kahlert C, Klupp F, Suarez-Carmona M, Suetterlin T, Brand K, Krauss J, Lasitschka F, Lerchl T, Luckner-Minden C, Ulrich A, Koch M, Weitz J, Schneider M, Buechler MW, Zitvogel L, Herrmann T, Benner A, Kunz C, Luecke S, Springfeld C, Grabe N, Falk CS, Jaeger D. Tumoral Immune Cell Exploitation in Colorectal Cancer Metastases Can Be Targeted Effectively by Anti-CCR5 Therapy in Cancer Patients. Cancer Cell. 2016 Apr 11;29(4):587-601. doi: 10.1016/j.ccell.2016.03.005. PMID 27070705